CLINICAL TRIAL: NCT07241689
Title: Effects of Protein Supplementation on 4 Weeks of Alternate-Day Fasting on Blood Parameters and Body Composition in Young Men
Brief Title: Effects of Protein Supplementation on 4 Weeks of Alternate-day Fasting on Fasting Blood Glucose, Resting Blood Pressure, and Body Composition in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2017-08-010
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight
Keywords: overweight; obesity; intermittent fasting; alternate-day fasting; body composition; muscle; fat; blood pressure; blood glucose; protein supplementation; weight loss
MeSH Terms: conditions — Obesity; Overweight; Intermittent Fasting; Platelet Glycoprotein IV Deficiency; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard ADF protocol of a small meal of their choice between 400-600 kcal on 12-2pm during fasting days
  Interventions: Other: No supplementation
- Protein (Experimental): ADF protocol of a small meal between 400-600 kcal including the protein supplement (125 kcal, 25 g protein) that is provided and with the remainder of the meal of their choice on 12-2pm during fasting days
  Interventions: Dietary Supplement: protein supplement

INTERVENTIONS:
Dietary Supplement: protein supplement — Protein supplement in the form of a whey protein powder containing 25 g of protein and 125 kcal that is provided during the fasting days
  Arms: Protein
Other: No supplementation — Standard ADF protocol of a small meal of their choice between 400-600 kcal during fasting days
  Arms: Control

SUMMARY:
The objectives of this study are to examine the effects of protein supplementation on 4 weeks of alternate-day fasting (ADF) on fasting blood glucose, resting blood pressure, and body composition in young Asian men with unhealthy body mass index ≥ 23 kg/m2.

To achieve the objective, 40 young men aged 21 to 35 years old will be recruited to participate in this study and complete a 4-week ADF programme. The fasting programme starts at 12 midnight and alternates between fasting and feeding days. Each fasting or feeding day is 24-hour in duration. On fasting days, no food and beverages are allowed except for ad libitum intake of plain water and/or other zero-calorie beverages, and a small meal between 400-600 kcal. In this study, participants would be randomly assigned to either the control or protein supplementation group (20 in each group). The control group will consume a small meal of their choice as long as it is between 400-600 kcal while the protein supplementation group will consume a small meal between 400-600 kcal that will include a protein supplement that would be provided (125 kcal, 25 g protein) and with the remainder of the meal of their choice. For both groups in this study, the small meal is to be consumed during 12 pm to 2 pm for standardisation to ensure consistency in total duration of fasting and feeding. The programme will end after 4 weeks (28 days) of continuous alternate-day fasting.

Fasting blood glucose, resting blood pressure and heart rate, body mass, height, and body composition will be measured before and after 4-week of ADF. In addition, these measurements, except body composition, will be repeated at the end of each week of ADF.

The research hypothesis are: 1) 4 weeks of ADF will reduce body mass via both fat and muscle loss, and improve health indices as measured by fasting blood glucose and resting blood pressure in young individuals with BMI greater than the desired healthy range, and 2) protein supplementation during fasting days will reduce muscle loss during loss of body mass.

DETAILED DESCRIPTION:
Methods Overview Participation in this study requires a total of 4 weeks of alternate-day fasting and 5 laboratory visits (sessions) spread over 5 weeks.

To participate in this study, participants will have to 1) sign the consent form, 2) complete a questionnaire which assesses their health with respect to the inclusion and exclusion criteria to ensure their safety and participation eligibility, 3) complete weekly questionnaire about their physical activity level, 4) complete 5 times of a health screening (measurement of resting blood pressure and heart rate, fasting blood sugar, body mass and height), 5) complete 2 occasions of body composition measurement, 6) complete 4 weeks of alternate-day fasting programme, and 7) complete 4 x 2-day dietary recalls for a total of 8 days of dietary recalls. Participants will also be required to consume a protein supplement on fasting days if assigned to the protein supplementation group.

Participants are required to:

1. follow the fasting programme as instructed including the protein supplementation if assigned (details given below),
2. abstain from taking medication (including traditional Chinese medicine) not previously declared unless when ill (participants are instructed to inform the investigators immediately if they fall ill during the study), hormones, steroids, and any supplements external to the study, including protein, vitamin and mineral supplements during the entire duration of the study,
3. maintain a consistent physical activity level throughout the entire duration of the study,
4. abstain from any physical activity except for activities of daily living for at least 48 hours prior to each session,
5. abstain from alcohol and caffeine for at least 24 hours prior to each session,
6. fast overnight for 10 hours before each session. In consideration of the fasting and to control for diurnal variation, all sessions will take place in the morning, and
7. abstain from all food and beverages during each session except for plain water that you may drink as much as you need.

Session 1: Consent, Questionnaires, Health Screening and Body Composition

Procedures involved:

1. Read and sign consent form if participating
2. Complete Subject Screening Questionnaire (to assess participants' health with respect to the inclusion and exclusion criteria to ensure their safety and participation eligibility)
3. Complete Global Physical Activity Questionnaire (GPAQ; to assess participants' physical activity level)
4. Answer questions related to health with respect to the inclusion and exclusion criteria
5. Have resting blood pressure and heart rate, body mass, and height measured
6. Have fasting blood sugar level measured using finger prick sampling
7. Undergo a direct segmental multi-frequency bioelectrical impedance analysis (DSM-BIA) to determine body composition
8. Collect the weekly supply of protein supplement in the form of a protein powder to be mixed with a beverage of their choice and to be consumed during the fasting days (see below) for participants assigned to the protein supplementation group.

Alternate-Day Fasting for 4 weeks (start within 1 week from session 1)

Procedures involved:

1. Programme starts at 12 midnight
2. Alternate between fasting and feeding days
3. Each fasting or feeding day is 24-hour in duration
4. On fasting days: no food and beverages except for ad libitum intake of plain water and/or other zero-calorie beverages, and a small meal between 400-600 kcal. In this study, participants would be randomly (by chance) assigned to either the standard or protein supplementation group. The standard group will consume a small meal of their choice as long as it is between 400-600 kcal while the protein supplementation group will consume a small meal between 400-600 kcal including the protein supplement (125 kcal, 25 g protein) that is provided and with the remainder of the meal of their choice.
5. For both groups in this study, this small meal is to be consumed during 12 pm to 2 pm for standardisation to ensure consistency in total duration of fasting and feeding. One must finish the protein supplement during this period of time if assigned to the protein supplementation group.
6. On feeding days: ad libitum eating except no alcohol and caffeine for at least 24 hours prior to sessions 2 to 4 if coinciding with the feeding days.
7. Programme ends after 4 weeks (28 days) of continuous alternate-day fasting

Sessions 2 to 4: Dietary Recalls, Health Screening and Questionnaire (at the end of each week of alternate-day fasting, ~1 hour for each session)

Procedures involved:

1. Complete a 2-day dietary recall on any 2 fasting days for the past week prior to each session
2. Have resting blood pressure and heart rate, body mass, and height measured
3. Have fasting blood sugar level measured using finger prick sampling
4. Complete Global Physical Activity Questionnaire (GPAQ)
5. Collect weekly supply of protein supplement if assigned to the protein supplementation group

Session 5: Dietary Recalls, Health Screening, Questionnaire and Body Composition (last session after 4 weeks of alternate-day fasting, ~1.5 hours)

Procedures involved:

1. Complete a 2-day dietary recall on any 2 fasting days for the past week prior to the session
2. Have resting blood pressure and heart rate, body mass, and height measured
3. Have fasting blood sugar level measured using finger prick sampling
4. Complete Global Physical Activity Questionnaire (GPAQ)
5. Undergo a direct segmental multi-frequency bioelectrical impedance analysis (DSM-BIA) to determine body composition

ELIGIBILITY:
Inclusion Criteria:

* Male
* 21 to 35 years old
* Do not smoke or use tobacco products (including shisha)
* Have a body mass index (BMI = body mass in kilograms divided by the square of height in metres) of 23 or greater

Exclusion Criteria:

One cannot participate in or will be released from this study if any of the following conditions or situations applies to them:

* Unable to adhere to requirements regarding physical activity and diet as stated in the methods
* Failed an exercise stress test
* Have any health condition(s) that would be made worse by fasting
* Taking long-term prescribed medication(s) for heart, blood (including blood glucose and blood pressure), lung (except controlled asthma), liver, kidney or joint condition(s)
* Taking other long-term prescribed medication (including traditional Chinese Medicine and other alternative medicine) that are known to affect any of the measurements in this study
* Allergic or intolerant to milk and soy (the protein supplement that participant may be required to consume, contains milk proteins and traces of soy lecithin and lactose)
* Have an artificial electrical implant such as a defibrillator or pacemaker

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Body mass | Start and end of 4-week intervention
  Body mass - a component of body composition.
Fat mass | Start and end of 4-week intervention
  A component of body composition. Total amount of fat mass.
Fat-free mass | Start and end of 4-week intervention
  A component of body composition. Total amount of fat-free mass, which is the total body mass excluding fat. It consists of primarily skeletal muscle mass, and also bone mass.
Skeletal muscle mass | Start and end of 4-week intervention
  A component of body composition. Total amount of skeletal muscle mass.
Appendicular fat-free mass | Start and end of 4-week intervention
  A component of body composition. Sum of skeletal muscle mass in the upper and lower limbs.
Percentage body fat | Start and end of 4-week intervention
  A component of body composition. Percentage of body mass that is made up of fat mass.
Visceral fat area | Start and end of 4-week intervention
  A component of body composition. Amount of visceral fat - a measurement of fat around abdominal organs.
Body mass index | Start and end of 4-week intervention
  A component of body composition. Computed from the measured body mass in kilograms divided by the square of height in metres.
Fat mass index | Start and end of 4-week intervention
  A component of body composition. Total fat mass in kilograms divided by square of height in metres.
Fat-free mass index | Start and end of 4-week intervention
  A component of body composition. Total fat-free mass in kilograms divided by square of height in metres.
Skeletal muscle mass index | Start and end of 4-week intervention
  A component of body composition. Total skeletal muscle mass divided by square of height in metres.
Appendicular fat-free mass index | Start and end of 4-week intervention
  A component of body composition. Total appendicular fat-free mass in kilograms divided by square of height in metres.

SECONDARY OUTCOMES:
Fasting blood glucose | Weekly from start to end of 4-week intervention
  Fasting blood glucose
Resting blood pressure | Weekly from start to end of 4-week intervention
  Resting blood pressure

OTHER OUTCOMES:
Hydration status | Start and end of 4-week intervention
  Intracellular water (litre)/extracellular water (litre). This ratio is a reflection of the hydration status in the body. Hydration status can affect the body composition measurements using bioelectrical impedance analysis.
Physical activity level | Weekly from start to end of 4-week intervention
  Weekly physical activity level estimated using Global Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Individual participant data (IPD) will be made available to qualified researchers upon request. To access the data, researchers must submit a formal request, which will be reviewed and approved by the data sharing committee. Data access will be granted for research purposes only and will require adherence to data use agreements and ethics guidelines.